CLINICAL TRIAL: NCT05389280
Title: Impact of Acute Kidney Injury on Sarcopenia and Frailty in Patients With Liver Cirrhosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kangbuk Samsung Hospital (Other)
Responsible Party: Principal Investigator, Won Sohn, Principal Investigator, Kangbuk Samsung Hospital
Other Study IDs: KBSMCLC2022
Record Dates: First submitted 2022-05-19; First posted 2022-05-25 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Cirrhosis; Kidney Injury; Sarcopenia; Frailty
MeSH Terms: conditions — Fibrosis; Sarcopenia; Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples Without DNA — Serum for testing NGAL, KIM-, and IL-18
  - Use a serum separator tube (SST) and allow samples to clot for 30 minutes at room temperature before centrifugation for 15 minutes at 1000 x g. Remove serum and assay immediately or aliquot and store samples at ≤ -20 °C. Avoid repeated freeze-thaw cycles.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this prospective observational study is to evaluate the impact of acute kidney injury on sarcopenia and frailty in patients with liver cirrhosis.

DETAILED DESCRIPTION:
The aim of this prospective study is to collect data on patients with liver cirrhosis and to investigate the impact of acute kidney injury on sarcopenia and frailty in patients with liver cirrhosis. If patients agree to participate in this clinical trial, the patients' data (such as age, sex, height, weight, nutrition status [RFH-NPT], history of medication, laboratory findings, endoscopic findings, and radiologic findings) will be collected in a research database. Renal injury was measured using conventional and novel serum biomarkers (serum creatinine, cystatin-C, neutrophil gelatinase-associated lipocalin, kidney injury molecule 1, and interleukin-18. Sarcopenia was evaluated using skeletal muscle index on abdominal computed tomography. Frailty was measured using Liver Frailty Index. The research database will be updated to include data on patients' disease outcomes and follow-up care.

ELIGIBILITY:
Inclusion Criteria:

* Liver cirrhosis
* aged over 20 years

Exclusion Criteria:

* serum creatinine >1.5 mg/dL
* on dialysis
* liver transplant

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with liver cirrhosis and serum creatinine <1.5 mg/dL
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-03-23 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Acute kidney injury | up to 24 weeks
  an increase in SCr of 0.3 mg/dL (26.4 µmoL/L) in <48 hours, or a 50% increase in SCr from a baseline within ≤3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Kangbuk Samsung Hospital, Seoul, South Korea